CLINICAL TRIAL: NCT02531334
Title: Effects of TA-65, a Telomerase Activator on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H14-278
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TA-65 (Experimental): TA-65 will be provided to volunteers for 12 weeks, two pills per day of 8 mg each
  Interventions: Dietary Supplement: TA-65
- Placebo (Placebo Comparator): Placebo will be provided to volunteers for 12 weeks, two pills per day of 8 mg each
  Interventions: Dietary Supplement: TA-65

INTERVENTIONS:
Dietary Supplement: TA-65 — 2 pills of TA-65 or placebo daily for 12 weeks. Subjects will be monitored weekly for side effects and every 4 weeks for compliance and safety monitoring. The whole intervention is a randomized double blind study for a duration of 27 weeks; 12 weeks for TA-65 or placebo allocated randomly and after a 3 week washout period, allocation to the alternate supplement TA-65 or placebo.

SUMMARY:
This study is being conducted to evaluate the efficacy of TA-65, a purified extract of Astragalus root, on insulin resistance, oxidative stress, and inflammation in individuals classified with metabolic syndrome.

DETAILED DESCRIPTION:
Short telomeres are strongly linked to increased risk of cardiovascular disease and diabetes, indications where tissue aging and senescence play significant roles. Shorter leukocyte telomere length has been linked to impaired glucose tolerance, Type 2 Diabetes, and coronary heart disease. Telomere length and telomerase activity have been shown to be significantly lower in CAD patients. Telomere length may play an important role in predicting cardiovascular disease and diabetes. TA-65 may not only ameliorate the symptoms associated with these disease states, but be a preventive measure as well.

In this study, the researchers will investigate whether telomerase activator (TA)-65 can also improve the metabolic dysregulations associated with metabolic syndrome including oxidative stress, inflammation, high blood pressure and dyslipidemias.

ELIGIBILITY:
Inclusion Criteria:

1. Age 32 to 70 years
2. Men and women
3. Proficiency in English
4. Postmenopausal women, or women of childbearing age (premenopausal) must be using some form of contraception or have had a hysterectomy
5. Classification of metabolic syndrome according to the Adult treatment panel (ATP) III criteria, meaning that individuals have 3 or more of the following characteristics:

   * Waist circumference >102 cm for men or > 88 cm for women
   * Triglycerides > 150 mg/d L
   * HDL cholesterol < 40 mg/dL for men or < 50 mg/dL for women
   * Blood pressure > 130/85 mm Hg or systolic ≥ 130 or diastolic ≥ 85*
   * Fasting blood glucose > 100 mg/dL *Or taking blood pressure medications

Exclusion Criteria:

1. Participants who do not fulfill the classification of metabolic syndrome, which means that they do not have 3 or more of the 5 characteristics previously mentioned
2. Participants with a body mass index (BMI) > 40 kg/m2
3. Current or past diagnosis of liver disease, renal disease, diabetes, cancer, stroke, heart disease, severe infectious disease, or autoimmune diseases (including but not limited to multiple sclerosis, lupus, and rheumatoid arthritis)
4. Women who are pregnant, lactating, or planning to become pregnant
5. Use of any glucose-lowering prescriptions or supplements, such as Sulfonylureas (Glucotrol, Amaryl, chlorpropamide, gliclazide, glimepiride, glipizide, glyburide), Thiazolidinediones (Avandia, ACTOS, rosiglitazone, pioglitazone), Meglitinides (Prandin, Starlix), Biguanides (Metformin), Alpha-glucosidase inhibitors (Precose, Glyset, acarbose, miglitol), Dipeptidyl peptidase (DPP)-4 inhibitors (Januvia, Onglyza, alogliptin, linagliptin, saxagliptin, sitagliptin), Glucagon-like peptide (GLP-1) antagonists (exenatide, liraglutide), Meglitinides (nateglinide, repaglinide), sodium glucose cotransporter (SGLT)-2 inhibitors (canagliflozin) or high dose chromium or cinnamon supplements
6. Use of immunosuppressants, including azathioprine, cyclophosphamide, basiliximab, cyclosporine, everolimus, daclizumab, infliximab, mercaptopurine, methotrexate, muromonab-cluster of differentiation3 (CD3), mycophenolate, pimecrolimus, rituximab, tacrolimus, sirolimus, prednisone, methylprednisone, dexamethasone, hydrocortisone (not topical), or prednisolone
7. Use of anticoagulants, including factor Xa inhibitors (rivaroxaban, apixaban), thrombin inhibitor (dabigatran), vitamin K antagonist (warfarin), heparin, low-molecular weight heparin, fondaparinux, or antiplatelets (aspirin, cilostazol, clopidogrel, dipyridamole, prasugrel, ticagrelor, ticlopidine)
8. Use of other categories of drugs, including methadone, Suboxone, monoamine oxidase (MAO) inhibitors, or lithium.
9. Use of any combination drug product containing any of the individual drugs listed above
10. Participants who have been consistently taking vitamin, mineral, or multivitamin supplements prior to recruitment may be admitted into the study if they plan to maintain their current supplement program. However, subjects may not participate if they begin taking a new supplement during the 27-week study period.
11. Fasting plasma triglycerides ≥ 500 mg/dL, glucose ≥ 126 mg/dL, or blood pressure > 145/100 mm Hg or systolic > 145 mm Hg or diastolic > 100 mm Hg

Ages: 32 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Plasma insulin | 27 weeks
  The supplement is expected to decrease insulin resistance in metabolic syndrome patients

SECONDARY OUTCOMES:
Plasma HDL cholesterol | 27 weeks
  The supplement is expected to increase plasma HDL cholesterol

OTHER OUTCOMES:
Blood pressure | 27 weeks
  The supplement is expected to decrease blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Fernandez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Result] Maubaret CG, Salpea KD, Jain A, Cooper JA, Hamsten A, Sanders J, Montgomery H, Neil A, Nair D, Humphries SE; HIFMECH consortium, Simon Broome Research Group. Telomeres are shorter in myocardial infarction patients compared to healthy subjects: correlation with environmental risk factors. J Mol Med (Berl). 2010 Aug;88(8):785-94. doi: 10.1007/s00109-010-0624-3. Epub 2010 Apr 11. PMID 20383691